CLINICAL TRIAL: NCT05733364
Title: Effect of 4 Weeks Supplementation of a Combination of Vitamin Bs and Taurine on Mental Performance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21.11.DAI
Record Dates: First submitted 2023-01-19; First posted 2023-02-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Healthy Working Adults
MeSH Terms: interventions — Taurine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, 2-arm, cross over trial. Participants will receive both the investigational product and placebo, each administered separately for a duration of 28 days, separated by a washout period of 28 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Product (Capsules with B vitamins & taurine) (Experimental): IP will be administered orally once daily in capsule form, ideally between conventional mealtimes (i.e., breakfast, lunch, supper).
  Interventions: Dietary Supplement: Capsules with B vitamins & taurine
- Microcrystalline cellulose placebo (Placebo Comparator): Placebo will be administered orally once daily in identical capsule form as the IP, ideally between conventional mealtimes (i.e., breakfast, lunch, supper).
  Interventions: Other: Microcrystalline cellulose placebo

INTERVENTIONS:
Dietary Supplement: Capsules with B vitamins & taurine — Administered orally in a span of 28 days between mealtimes
  Arms: Investigational Product (Capsules with B vitamins & taurine)
Other: Microcrystalline cellulose placebo — Administered orally in a span of 28 days between mealtimes
  Arms: Microcrystalline cellulose placebo

SUMMARY:
To evaluate the efficacy of the intervention in improving Motivation.

To evaluate the efficacy of the intervention in improving Fatigue, Motivation/Vigor, Focus/Sustained Attention and blood levels of B vitamins and taurine.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, aged 25-40 years, inclusive, at enrolment.
* Healthy as per site physician/investigator medical assessment based on medical history and physical examination.
* Body mass index (BMI) between 18.5 to 27.5 kg/m².
* Able to understand and provide signed informed consent prior to study enrolment.
* Willing and able to comply with the requirements for participation in this study.
* Day time workers who work ≥ 8 and ≤ 12 hours per day, and ≤ 60 hours per week.

Exclusion Criteria:

* Any significant ongoing or past medical (including celiac disease, obstructive sleep apnea, restless leg syndrome) and/or psychiatric condition, which in the opinion of the site physician/investigator may compromise participant wellbeing/safety, impede participant compliance with study procedures, or ability to complete the study.
* Any clinically significant abnormality detected by the site physician/investigator during physical examination conducted at screening.
* Participants with reported intermediate visual acuity less than 20/25 and without correction.
* Known history of allergy to the ingredients in the investigational products.
* Participants that have taken part in another interventional clinical trial within the last 3 months.
* Current regular smoker (regularity defined ≥2 cigarettes per week).
* Pregnant, lactating, or intending to conceive during the clinical trial.
* Use of chronic over the counter or prescription medicines that may affect cognitive and physical functioning within 30 days or 5 half-lives prior to enrolment e.g., antidepressants, anxiolytics, antihistamines, narcotic analgesics.
* Alcohol consumption above daily recommended alcohol intake for men (2 drinks = 24 g/day) and women (1 drink = 12 g/day) (assessed by self-report; local guidelines)
* Caffeine consumption above recommended caffeine daily consumption, defined as > 400 mg/day (approximately 4 cups of coffee), and evaluated using the Caffeine Consumption Questionnaire.
* Consumption of energy drinks containing Taurine and/or Vitamin Bs within 21 days prior to enrolment
* Use of vitamin Bs and/or Whey protein and/or amino acid supplements within 30 days of enrolment.
* Presence of sleep disorders (evaluated using the global sleep assessment questionnaire (GSAQ))
* Performing shift work or trans-meridian travel within 10 days of enrolment

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the intervention in improving Motivation | 28 days
  The mean change from baseline to day 28 of product intake across sessions in the Monetary Incentivized Delay Task (MIDT). Assessment will be recorded as number of success over total in fraction or in %

SECONDARY OUTCOMES:
To evaluate the efficacy of the intervention in improving Fatigue. | 28 days
  Profile of Mood States short-form 2 (POMS-SF 2): change in self-reported levels of fatigue/inertia. Assessment will be recorded as score in arbitrary units (A.U.)
To evaluate the efficacy of the intervention in improving Fatigue. | 28 days
  NASA Task Load Index (NASA-TLX): changes in self-reported levels of perceived mental, physical, and temporal demands, self-perceived overall performance, levels of perceived effort exertion and levels of frustration. Assessment will be recorded as score in arbitrary units (A.U.)
To evaluate the efficacy of the intervention in improving Focus | 28 days
  Capacity to sustain high levels of attention: Psychomotor Vigilance Task. Assessment will be recorded as total number of lapses in absolute number.
To evaluate the efficacy of the intervention in improving Vigor. | 28 days
  POMS-SF 2: change in self-reported levels of vigor. Assessment will be recorded as score in arbitrary units (A.U.)
To evaluate the efficacy of the intervention in improving Focus | 28 days
  Capacity to sustain high levels of attention: Psychomotor Vigilance Task. Assessment will be recorded as reaction time in milisecond (ms)
To evaluate the efficacy of the intervention in improving Motivation | 28 days
  The mean change from baseline to day 28 of product intake across sessions in the Monetary Incentivized Delay Task (MIDT). Assessment will be recorded as effort or force in kilogram-force (kgf)
To evaluate the efficacy of the intervention in improving Vigor. | 28 days
  Self-reported motivation with the Global Motivation Scale: changes in intrinsic motivation, extrinsic motivation, and amotivation. Assessment will be recorded as score in arbitrary units (A.U.)

OTHER OUTCOMES:
To evaluate the effect of the intervention on blood levels of vitamins B6 & B9 | 28 days
  Change in level of vitamins B6 & B9 in blood at baseline and Day 28 of each administration period. Assessment will be recorded in microgram per litre (µg/L).
To evaluate the effect of the intervention on blood levels of vitamins B12 | 28 days
  Change in level of vitamin B12 in blood at baseline and Day 28 of each administration period. Assessment will be recorded in nanograms per litre (ng/L).
To evaluate the effect of the intervention on blood levels of taurine | 28 days
  Change in level of taurine in blood at baseline and Day 28 of each administration period. Assessment will be recorded in micromoles per litre (µmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Veeda M Anlacan, MD, Principal Investigator — University of the Philippines
Locations (1):
- Philippine General Hospital, Philippines, Philippines

IPD SHARING:
Plan to Share IPD: Undecided